CLINICAL TRIAL: NCT00164723
Title: Endoscopic Evaluation of the Incidence and Etiology of Lower Gastrointestinal Bleeding in Patients Presenting With Melena
Brief Title: Endoscopic Evaluation of Lower Gastrointestinal Bleeding (GIB) in Patients Presenting With Melena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CE_GIB
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2011-01

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Capsule Endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NSAID (Other): patients taking NSAID will undergo capsule endoscopy
  Interventions: Procedure: Capsule endoscopy
- Aspirin (Other): patients taking Aspirin will undergo capsule endoscopy
  Interventions: Procedure: Capsule endoscopy
- Non-user (Other): patients didn't take NSAID or ASA will undergo capsule endoscopy
  Interventions: Procedure: Capsule endoscopy

INTERVENTIONS:
Procedure: Capsule endoscopy — Capsule endoscopy and colonoscopy

SUMMARY:
To evaluate the incidence and etiology of small bowel or large bowel bleeding in patients presenting with melena.

DETAILED DESCRIPTION:
Although tarry stool is a common feature of peptic ulcer bleeding, it can also be a manifestation of lower gastrointestinal (GI) bleeding. Examples include colonic cancer, small bowel tumors, and small or large bowel ulcers induced by aspirin or painkillers (NSAIDs). However, clinicians are often misled by the finding of peptic ulcers as the source of GI bleeding. It is not uncommon to detect peptic ulcers incidentally but the source of bleeding is actually in the lower GI tract (e.g. NSAID- or aspirin-induced small or large bowel bleeding ulcers, small bowel tumors, or colorectal cancer). Delay in diagnosis of lower GI bleeding often leads to serious consequences.

The preferred investigations for lower GI bleeding are colonoscopy plus video capsule endoscopy. Colonoscopy has been the gold standard for the diagnosis of colonic bleeding. The risk of colonoscopy-induced complications such as bleeding or perforation is less than 1 in 3500. Video capsule endoscopy is a non-invasive, safe and accurate technology that has been approved by the FDA for investigation of small bowel diseases. The video capsule is an 11x 26mm capsule that encases a digital camera, light-emitting diodes, batteries, and a transmitter. The patient needs to swallow the video capsule after an overnight fast and wear a recording device for eight hours. Images are taken twice-per-second and transmitted to the recording device. Oral feeding can be resumed after four hours. There is no restriction to daily activities. The swallowed capsule will be expelled naturally after 5 to 12 hours virtually in all patients. The risk of capsule retention is very low and only occurs in patients with severe small bowel stricture.

This study aims to assess the incidence and etiology of lower GI bleeding in patients presenting with tarry stool. The result will provide important information about the magnitude of the problem of lower GI bleeding that will improve our patient care.

ELIGIBILITY:
Consecutive patients with a clinical diagnosis of upper gastrointestinal bleeding will be enrolled if they meet all of the following criteria:

1. Presence of melena or melena concomitant with PR bleeding;
2. Gastroscopic findings not accountable for the upper GI bleeding including: (i) clean base ulcers /erosions (refer to User Groups below) without high-risk stigmata, fresh or altered blood but can have grade A or B esophagitis concomitantly ; and (ii) meet the criteria of either the User groups or Non-user group as below

   User Groups Definition: Patients who used any dose of NSAIDs or aspirin via oral or systemic (intramuscular, Per rectal) route within 2 weeks prior to the onset of upper GI bleeding NSAID group: Clean base gastric or duodenal ulcer is required (i.e., patients with normal finding or erosions alone on endoscopy will not be eligible) Aspirin group: Either an ulcer or multiple (>5) erosions found on endoscopy

   Non-user group

   Definition :
   1. No continuous use of NSAIDs or aspirin for more than 1 week within the past 3 Months and patients who had not been exposed to NSAIDs, aspirin, or unknown drugs ≥ 4 weeks prior to GI bleed;
   2. Clean base gastric or duodenal ulcer is required (i.e., patients with normal finding or erosions alone on OGD will not be eligible)
3. Age ³18;
4. Willing to meet the capsule endoscopy procedure requirements, and have provided written informed consent prior to admission to this study.
5. Concomitant clean base GU and DU can be recruited

Exclusion criteria

The presence of any of the following will exclude a subject from study enrollment:

1. Hematemesis as the presenting symptom;
2. Gastroscopic findings accountable for the bleeding episode (i.e., presence of blood in the stomach, ulcers showing high-risk bleeding stigmata, bleeding gastroesophageal varices, Mallory-Weiss tear showing bleeding stigmata, portohypertensive gastropathy);
3. Gastroscopic findings are normal.
4. Uncontrolled bleeding requiring emergency surgery or mesenteric angiography;
5. Has cardiac pacemaker or other electromedical implant;
6. Is expected to undergo MRI examination or be in the vicinity of powerful electromagnetic fields between ingesting the capsule and its excretion;
7. Active malignancy or history of a malignancy within 5 years prior to enrollment;
8. Previous gastric surgery;
9. Known or suspected complete or partial stenosis of the small intestine;
10. Established delayed gastric emptying or diabetic gastroparesis;
11. Known inflammatory bowel disease;
12. Use of misoprostol within the 2 weeks prior to admission;
13. Concomitant use of NSAIDs and aspirin;
14. Currently taking anticoagulants or lithium;
15. Has a swallowing disorder that precludes safe ingestion of the capsule;
16. Pregnancy;
17. History of clinically significant substance abuse, drug addiction or a history of chronic ingestion of more than two alcoholic drinks per day;
18. Any mental or physical condition, which precludes compliance with study and/or device instructions;
19. Received any investigational medication within 30 days prior to the treatment period;
20. Currently participating in another clinical study that may affect the results of this study.
21. Ulcer > 2cm
22. clean base ulcer with grade C or D esophagitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of capsule endoscopy as the primary investigation for small bowel after negative esophagogastroduodenoscopy | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL Chan, MD, Principal Investigator — CUHK
Locations (1):
- Endoscopy Center in Prince of Wales Hospital, Hong Kong (sar), China